CLINICAL TRIAL: NCT01291264
Title: Evaluation of Abbott RealTime CT/NG for the Detection of Chlamydia Trachomatis [CT] & Neisseria Gonorrhoeae [NG] From the Pharynx, Rectum & Urethra of Men Who Have Sex With Men [MSM]
Brief Title: Use of Abbott RealTime CT/NG to Detect Chlamydia Trachomatis [CT] & Neisseria Gonorrhoeae [NG] in Men Who Have Sex With Men [MSM]
Status: Terminated | Type: Observational
Why Stopped: Abbott Molecular stopped funding of study
Sponsor: University of California, San Francisco (Other)
Collaborators: Abbott Molecular (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-04134
Record Dates: First submitted 2011-02-01; First posted 2011-02-08 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Chlamydia Infection; Gonococcal Infection; Sexually Transmitted Diseases
Keywords: Chlamydia trachomatis; Neisseria gonorrhoeae; Sexually Transmitted Diseases
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — clinician-collected rectal and pharyngeal swabs along with FCUs
Oversight: Data Monitoring Committee: No

SUMMARY:
Julius Schachter, PhD, (Department of Laboratory Medicine, University of California, San Francisco) and Susan S. Philip, MD MPH (Department of Medicine, University of California, San Francisco) are conducting a study to evaluate the Abbott RealTime CT/NG polymerase chain reaction [PCR] assay (which is a nucleic acid amplification test [NAAT]) for detecting two sexually transmitted bacteria, Chlamydia trachomatis [CT] and Neisseria gonorrhoeae [NG], using urine samples and swabs from the throat and rectum of men who have sex with men [MSM]. Using this test on these swabs is experimental because it has not been approved by the Food & Drug Administration.

DETAILED DESCRIPTION:
For each subject enrolled in the study, the following clinical data information will be obtained: 1) reason for exam, 2) subject's signs and symptoms and 3) clinical assessment.

For each subject enrolled in the study, two clinician-collected pharyngeal swabs, two clinician-collected rectal swabs, and a first catch urine specimen (approximately 25 ml) will be obtained. The collection order of the clinician-collected swabs will be randomized.

Two pharyngeal swabs will be tested at the research laboratory using: 1) APTIMA COMBO 2® [AC2](Gen-Probe Inc, San Diego, CA); and 2) Abbott RealTime CT/NG [RealTime](Abbott Molecular, Des Plains, IL). Two rectal swabs will be tested at the research laboratory using: 1) AC2; and 2) RealTime.

A first-catch urine [FCU] specimen will be split out at San Francisco Department of Public Health laboratory and sent to the Chlamydia Research Laboratory for analysis using: 1)AC2; and 2) RealTime.

All NAAT specimens are collected in the manufacturer's recommended NAAT transport medium. After specimen processing, samples will be frozen at -70ºC for discrepant analysis.

ELIGIBILITY:
Inclusion Criteria:

* A subject must be MSM. Subjects must provide verbal consent, must be able to submit all required specimens and must not have urinated within 1 hr prior to providing a study urine specimen.

Exclusion Criteria:

* Subjects are excluded if they do not have sex with men, refuse to give verbal consent or refuse to allow such consent to be documented in their chart, are unable to provide all required specimens and minimum specimen volume, have been on antibiotic therapy within the last 21 days, have urinated within 1 hr prior to submitting study specimens, and have already been evaluated as part of this trial. Subjects will be excluded if specimens are mishandled or inappropriately stored.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men who have sex with men (MSM) voluntarily presenting at the City STD clinic.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Schachter, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - SF City Clinic, San Francisco, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Background] Johnson RE, Newhall WJ, Papp JR, Knapp JS, Black CM, Gift TL, Steece R, Markowitz LE, Devine OJ, Walsh CM, Wang S, Gunter DC, Irwin KL, DeLisle S, Berman SM. Screening tests to detect Chlamydia trachomatis and Neisseria gonorrhoeae infections--2002. MMWR Recomm Rep. 2002 Oct 18;51(RR-15):1-38; quiz CE1-4. PMID 12418541
- [Background] Workowski KA, Berman S; Centers for Disease Control and Prevention (CDC). Sexually transmitted diseases treatment guidelines, 2010. MMWR Recomm Rep. 2010 Dec 17;59(RR-12):1-110. PMID 21160459
- [Background] Page-Shafer K, Graves A, Kent C, Balls JE, Zapitz VM, Klausner JD. Increased sensitivity of DNA amplification testing for the detection of pharyngeal gonorrhea in men who have sex with men. Clin Infect Dis. 2002 Jan 15;34(2):173-6. doi: 10.1086/338236. Epub 2001 Dec 7. PMID 11740704
- [Background] Van Der Pol B, Ferrero DV, Buck-Barrington L, Hook E 3rd, Lenderman C, Quinn T, Gaydos CA, Lovchik J, Schachter J, Moncada J, Hall G, Tuohy MJ, Jones RB. Multicenter evaluation of the BDProbeTec ET System for detection of Chlamydia trachomatis and Neisseria gonorrhoeae in urine specimens, female endocervical swabs, and male urethral swabs. J Clin Microbiol. 2001 Mar;39(3):1008-16. doi: 10.1128/JCM.39.3.1008-1016.2001. PMID 11230419
- [Background] Ciemins EL, Flood J, Kent CK, Shaw H, Rowniak S, Moncada J, Klausner JD, Schachter J. Reexamining the prevalence of Chlamydia trachomatis infection among gay men with urethritis: implications for STD policy and HIV prevention activities. Sex Transm Dis. 2000 May;27(5):249-51. doi: 10.1097/00007435-200005000-00002. PMID 10821595
- [Background] Rompalo AM, Price CB, Roberts PL, Stamm WE. Potential value of rectal-screening cultures for Chlamydia trachomatis in homosexual men. J Infect Dis. 1986 May;153(5):888-92. doi: 10.1093/infdis/153.5.888. PMID 3084665
- [Background] Chernesky MA, Martin DH, Hook EW, Willis D, Jordan J, Wang S, Lane JR, Fuller D, Schachter J. Ability of new APTIMA CT and APTIMA GC assays to detect Chlamydia trachomatis and Neisseria gonorrhoeae in male urine and urethral swabs. J Clin Microbiol. 2005 Jan;43(1):127-31. doi: 10.1128/JCM.43.1.127-131.2005. PMID 15634960
- [Background] Schachter J, Moncada J, Liska S, Shayevich C, Klausner JD. Nucleic acid amplification tests in the diagnosis of chlamydial and gonococcal infections of the oropharynx and rectum in men who have sex with men. Sex Transm Dis. 2008 Jul;35(7):637-42. doi: 10.1097/OLQ.0b013e31817bdd7e. PMID 18520976
- [Background] Kent CK, Chaw JK, Wong W, Liska S, Gibson S, Hubbard G, Klausner JD. Prevalence of rectal, urethral, and pharyngeal chlamydia and gonorrhea detected in 2 clinical settings among men who have sex with men: San Francisco, California, 2003. Clin Infect Dis. 2005 Jul 1;41(1):67-74. doi: 10.1086/430704. Epub 2005 May 26. PMID 15937765
- [Background] Laboratory Diagnostic Testing for Chlamydia trachomatis and Neisseria gonorrhoeae. American Public Health Laboratories/Center for Disease Control & Prevention Panel Summary Reports. January 2009. Internet. Accessed 8 November 2010. http://www.aphl.org/aphlprograms/infectious/std/Documents/CTGCLabGuidelinesMeetingReport.pdf
- [Background] Moncada J, Schachter J, Liska S, Shayevich C, Klausner JD. Evaluation of self-collected glans and rectal swabs from men who have sex with men for detection of Chlamydia trachomatis and Neisseria gonorrhoeae by use of nucleic acid amplification tests. J Clin Microbiol. 2009 Jun;47(6):1657-62. doi: 10.1128/JCM.02269-08. Epub 2009 Apr 15. PMID 19369445
- [Background] Gaydos CA, Cartwright CP, Colaninno P, Welsch J, Holden J, Ho SY, Webb EM, Anderson C, Bertuzis R, Zhang L, Miller T, Leckie G, Abravaya K, Robinson J. Performance of the Abbott RealTime CT/NG for detection of Chlamydia trachomatis and Neisseria gonorrhoeae. J Clin Microbiol. 2010 Sep;48(9):3236-43. doi: 10.1128/JCM.01019-10. Epub 2010 Jul 28. PMID 20668135

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates were 06/06/12 to 09/19/12. Study was done at the San Francisco City STD Clinic.
Groups:
- Men Who Have Sex With Men: The study population consisted of asymptomatic and symptomatic MSM that could provide approximately 25 ml of first catch urine (FCU), and two clinician-collected pharyngeal and rectal swabs.
Period: Overall Study
Arm/Group | Men Who Have Sex With Men
Started | 260
Completed | 260
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Men who have sex with men
Arm/Group | Men Who Have Sex With Men
Number analyzed (Participants) | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 260
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 260

OUTCOME MEASURES:

1. Primary Outcome: Subject's Infected-status as Determined by the Nucleic Acid Amplification Assays Performed.
Description: This is a single-point prevalence assessment done when subjects present at the STD clinic for routine STD screening. Subjects are not followed beyond the clinic visit.
Time Frame: 1 day - (At clinic visit)
Population: per protocol
Measure: Number; unit: Positive test result
Arm/Group | Men Who Have Sex With Men
Number analyzed (Participants) | 260
Positive test result
  Oropharynx tested by RealTime for NG | 11
  Oropharynx tested by AC2 for NG | 12
  Rectum tested by RealTime for NG | 16
  Rectum tested by AC2 for NG | 20
  FCU tested by RealTime for NG | 11
  FCU tested by AC2 for NG | 12
  Oropharynx tested by RealTime for CT | 0
  Oropharynx tested by AC2 for CT | 0
  Rectum tested by RealTime for CT | 17
  Rectum tested by AC2 for CT | 17
  FCU tested by RealTime for CT | 9
  FCU tested by AC2 for CT | 8

ADVERSE EVENTS:
Arm/Group | Men Who Have Sex With Men
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Our limitations are small number of subjects enrolled due to early termination of the study and we had no pharyngeal CT infections.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No